CLINICAL TRIAL: NCT02677324
Title: Phase II Study of ABT-199 (GDC-199) In Patients With Relapsed Or Refractory Waldenström Macroglobulinemia
Brief Title: Study of ABT-199 (GDC-199) In Patients With Relapsed Or Refractory Waldenström Macroglobulinemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Principal Investigator, Jorge J. Castillo, MD, Jorge J. Castillo, MD, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-491; A15-751 (Other: AbbVie Inc)
Record Dates: First submitted 2016-01-14; First posted 2016-02-09 (Estimated); Results first posted 2021-05-11 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-04

CONDITIONS: Waldenstrom Macroglobulinemia
Keywords: Waldenstrom Macroglobulinemia; WM
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ABT199 (Experimental): ABT199 will be administered daily, with 28 consecutive days defined as a treatment cycle for a maximum for 26 cycles
  Interventions: Drug: ABT199

INTERVENTIONS:
Drug: ABT199 — Oral BCL-2 antagonist
  Other Names: Venetoclax

SUMMARY:
This research study is studying a targeted therapy as a possible treatment for relapsed or refractory Waldenstrom's Macroglobulinemia (WM). This study is using the study intervention ABT-199.

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. ABT-199 is a pill that blocks BCL-2, a protein that is important for the survival of WM cells.

The purpose of this research study is to evaluate how well the study drug works and the safety of ABT-199 as a single agent in participants with WM that has come back or has shown no response to previous treatment.

The FDA (the U.S. Food and Drug Administration) has not approved ABT-199 as a treatment for any disease.

ELIGIBILITY:
Inclusion Criteria:

* Clinicopathological diagnosis of Waldenstrom's Macroglobulinemia and meeting criteria for treatment using consensus panel criteria from the Second International Workshop on Waldenstrom's macroglobulinemia (Owen 2003; Kyle 2003).
* Measurable disease, defined as presence of serum immunoglobulin M (IgM) with a minimum IgM level of > 2 times the upper limit of normal of each institution is required.
* Have received at least one prior therapy for WM.
* Age ≥ 18 years.
* ECOG performance status <2 (see Appendix A).
* Participants must have normal organ and marrow function (growth factors cannot be given prophylactically to establish eligibility) as defined below:

  * Absolute neutrophil count > 1,000/mm3
  * Platelets > 50,000/mm3
  * Hemoglobin > 8 g/dL
  * Total bilirubin ≤ 1.5 mg/dL or < 2 mg/dL if attributable to hepatic infiltration by neoplastic disease
  * AST (SGOT) and ALT (SGPT) < 2.5X the institutional upper limit of normal
  * Creatinine clearance ≥50 ml/min
* Not on any active therapy for other malignancies with the exception of topical therapies for basal cell or squamous cell cancers of the skin.
* Females of childbearing potential (FCBP) must agree to use two reliable forms of contraception simultaneously or have or will have complete abstinence from heterosexual intercourse during the following time periods related to this study: 1) while participating in the study; and 2) for at least 28 days after discontinuation from the study. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. FCBP must be referred to a qualified provider of contraceptive methods if needed.
* Able to adhere to the study visit schedule and other protocol requirements.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, uncontrolled intercurrent illness, or psychiatric illness/social condition that would prevent the participant from signing the informed consent form.
* Concurrent use of any other anti-cancer agents or treatments or any other study agents.
* Prior exposure to ABT-199 or BCL2 inhibitors.
* Prior or ongoing clinically significant illness, medical condition, surgical history, physical finding, ECG finding, or laboratory abnormality that, in the investigator's opinion, could affect the safety of the patient, including symptomatic hyperviscosity; alter the absorption, distribution, metabolism or excretion of ABT-199; or impair the assessment of study results.
* Grade > 2 toxicity (other than alopecia) continuing from prior anti-cancer therapy.
* Known CNS lymphoma.
* Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening.
* New York Heart Association classification III or IV heart failure.
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel, ulcerative colitis, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction.
* Known history of Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), and/or Hepatitis C Virus (HCV) infection.
* Lactating or pregnant women.
* Inability to swallow tablets.
* History of non-compliance to medical regimens.
* Unwilling or unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-05-09 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2022-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge J Castillo, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - City of Hope National Medical Center, Duarte, California
  - Stanford University, Palo Alto, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Weill Cornell Medical College, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Castillo JJ, Guijosa A, Allan JN, Siddiqi T, Advani RH, Flynn CA, Meid K, Budano N, Nguyen J, Ramirez-Gamero A, Tsakmaklis N, Hunter ZR, Patterson CJ, Treon SP, Sarosiek S. Long-term follow-up of venetoclax monotherapy in previously treated patients with Waldenstrom macroglobulinemia. Blood Adv. 2025 Oct 14;9(19):4842-4847. doi: 10.1182/bloodadvances.2025016890. PMID 40674749
- [Derived] Castillo JJ, Allan JN, Siddiqi T, Advani RH, Meid K, Leventoff C, White TP, Flynn CA, Sarosiek S, Branagan AR, Demos MG, Guerrera ML, Kofides A, Liu X, Munshi M, Tsakmaklis N, Xu L, Yang G, Patterson CJ, Hunter ZR, Davids MS, Furman RR, Treon SP. Venetoclax in Previously Treated Waldenstrom Macroglobulinemia. J Clin Oncol. 2022 Jan 1;40(1):63-71. doi: 10.1200/JCO.21.01194. Epub 2021 Nov 18. PMID 34793256

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ABT199
Started | 33
Completed | 21
Not Completed | 12
Not completed — Disease Progression | 6
Not completed — Inability to Swallow pills | 1
Not completed — Non-compliance | 1
Not completed — Lack of Efficacy | 1
Not completed — Medical insurance coverage | 1
Not completed — Adverse Event | 1
Not completed — IgM Myeloma diagnosis | 1

BASELINE CHARACTERISTICS:
Arm/Group | ABT199
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 19
Age, Continuous [Median (Full Range); unit: years] | 66 [39 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 30
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 33
MYD88 Mutation [Count of Participants; unit: Participants] | 32
CXCR4 Mutation [Count of Participants; unit: Participants] | 17

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall Response Rate= Minor response (>25%-50% reduction in serum IgM from baseline) + Partial Response (>50-90% reduction in serum IgM from baseline) + Very Good Partial Response (>90% reduction in serum IgM from baseline) + Complete Response (resolution of all symptoms, normalization of serum IgM with disappearance of IgM paraprotein, resolution of any adenopathy or splenomegaly).
Time Frame: 2 years
Population: 1 participant was censored from the response analysis after it was determined that he had IgM Myeloma rather than Waldenstrom's macroglobulinemia.
Measure: Count of Participants; unit: Participants
Arm/Group | ABT199
Number analyzed (Participants) | 32
Participants | 26

2. Secondary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0
Description: Number of participants who experienced an adverse event while on ABT-199
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | ABT199
Number analyzed (Participants) | 33
Participants | 33

3. Secondary Outcome: Number of Participants With Complete Response
Description: A complete response is defined as having resolution of WM related symptoms, normalization of serum IgM levels with complete disappearance of IgM paraprotein by immunofixation, and resolution of any adenopathy or splenomegaly.
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ABT199
Number analyzed (Participants) | 32
Participants | 0

4. Secondary Outcome: Number of Participants With Very Good Partial Response
Description: Very Good Partial Response (VGPR): is defined as ≥90% reduction in serum IgM levels, or normalization of serum IgM levels.
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ABT199
Number analyzed (Participants) | 32
Participants | 6

5. Secondary Outcome: Number of Participants With Partial Response
Description: Partial response (PR) is defined as achieving a ≥50% reduction in serum IgM levels.
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ABT199
Number analyzed (Participants) | 32
Participants | 19

6. Secondary Outcome: Number of Participants With Minor Response
Description: Minor Response (MR): A minor response (MR) is defined 25-49% reduction in serum IgM levels.
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ABT199
Number analyzed (Participants) | 32
Participants | 1

7. Secondary Outcome: Number of Participants With Stable Disease
Description: Stable disease is defined as having <25% increase in serum IgM levels and <25% reduction in serum IgM levels
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ABT199
Number analyzed (Participants) | 32
Participants | 2

8. Secondary Outcome: Progression Free Survival
Description: Amount of time following ABT-199 administration until >25% increase in serum IgM
Time Frame: 4 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ABT199
Number analyzed (Participants) | 32
months | 31.5 [26.6 to 38.6]

9. Secondary Outcome: Overall Response Rate Among CXCR4 Mutated Participants
Description: Overall Response Rate for participants who tested positive for a CXCR4 mutation= Minor response (>25%-50% reduction in serum IgM from baseline) + Partial Response (>50-90% reduction in serum IgM from baseline) + Very Good Partial Response (>90% reduction in serum IgM from baseline) + Complete Response (resolution of all symptoms, normalization of serum IgM with disappearance of IgM paraprotein, resolution of any adenopathy or splenomegaly).
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Groups:
- CXCR4 Mutated Participants: Participants with the CXCR4 mutation detected at baseline bone marrow assessment
Arm/Group | CXCR4 Mutated Participants
Number analyzed (Participants) | 17
Participants | 14

10. Secondary Outcome: Overall Response Rate Among Participants Without CXCR4 Mutations
Description: Overall Response Rate in participants who tested negative for a CXCR4 mutation= Minor response (>25%-50% reduction in serum IgM from baseline) + Partial Response (>50-90% reduction in serum IgM from baseline) + Very Good Partial Response (>90% reduction in serum IgM from baseline) + Complete Response (resolution of all symptoms, normalization of serum IgM with disappearance of IgM paraprotein, resolution of any adenopathy or splenomegaly).
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Groups:
- CXCR4 Wild-Type Participants: Participants who tested negative for a CXCR4 mutation at their baseline bone marrow assessment
Arm/Group | CXCR4 Wild-Type Participants
Number analyzed (Participants) | 15
Participants | 13

ADVERSE EVENTS:
Time Frame: Adverse events were collected from starting ABT-199, through study therapy, and up to 30 days after the last dose of ABT-199, for up to 2.5 years.
Arm/Group | ABT199
All-Cause Mortality (participants affected / at risk) | 0/33
Serious Adverse Events (participants affected / at risk) | 13/33
Other Adverse Events (participants affected / at risk) | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABT199 (N=33)
Upper Respiratory Infection (Infections and infestations) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Sepsis due to Pneumonia (Infections and infestations) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Laboratory tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Renal calculi (Renal and urinary disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Rectal bleeding (Gastrointestinal disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABT199 (N=33)
Fatigue (General disorders) | 23 (23)
Fever (General disorders) | 8 (8)
Pain (General disorders) | 6 (6)
Edema limbs (General disorders) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (9)
Non-cardiac chest pain (General disorders) | 4 (4)
Chills (General disorders) | 3 (3)
Dizziness (General disorders) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 11 (11)
Upper respiratory infection (Infections and infestations) | 15 (15)
Sinusitis (Infections and infestations) | 6 (6)
Urinary tract infection (Infections and infestations) | 4 (4)
Rash not otherwise specified (Skin and subcutaneous tissue disorders) | 10 (10)
Bruising (Injury, poisoning and procedural complications) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 2 (2)
Neutrophil count decreased (Investigations) | 22 (22)
Platelet count decreased (Investigations) | 13 (13)
Lymphocyte count decreased (Investigations) | 9 (9)
White blood cell decreased (Investigations) | 8 (8)
Aspartate aminotransferase increased (Investigations) | 5 (5)
Weight loss (Investigations) | 4 (4)
Alkaline phosphatase increased (Investigations) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 7 (7)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 6 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 9 (9)
Dizziness (Nervous system disorders) | 8 (8)
Headache (Nervous system disorders) | 7 (7)
Paresthesia (Nervous system disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 8 (8)
Depression (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 15 (15)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (12)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pruritis (Skin and subcutaneous tissue disorders) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertension (Vascular disorders) | 5 (5)
Hypotension (Vascular disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 18 (18)
Palpitations (Cardiac disorders) | 5 (5)
Sinus bradycardia (Cardiac disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Ventricular arrhythmia (Cardiac disorders) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 2 (2)
Blurred vision (Eye disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 20 (20)
Nausea (Gastrointestinal disorders) | 15 (15)
Constipation (Gastrointestinal disorders) | 8 (8)
Abdominal pain (Gastrointestinal disorders) | 7 (7)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 4 (4)
Bloating (Gastrointestinal disorders) | 3 (3)
Flatulence (Gastrointestinal disorders) | 3 (3)
Mucositis oral (Gastrointestinal disorders) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-18): https://cdn.clinicaltrials.gov/large-docs/24/NCT02677324/Prot_SAP_000.pdf